CLINICAL TRIAL: NCT04260256
Title: A Pilot Study of Using [18F]F AraG PET Imaging to Evaluate the Immunological Response to Checkpoint Inhibitor Therapy (CkIT) in Patients With Advanced Solid Tumors
Brief Title: A Study Using [18F]F AraG PET to Evaluate Response to Checkpoint Inhibitor Therapy(CkIT) in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Collaborators: Stanford University (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 53563; NCT05219981 (obsolete NCT alias)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Correlate Tracer Uptake to TCell Tumor Infiltration & CkIT Benefit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: [18F]F-AraG — [18F]F AraG injection and PET Scan Two tumor biopsies of single lesion
  Other Names: VisAcT

SUMMARY:
In this study, patients with advanced solid tumors will undergo [18F]F AraG PET/CT imaging to assess for changes in tracer uptake following treatment with CkIT.

DETAILED DESCRIPTION:
Up to 40 patients will be recruited to participate in this study. Two (2) target lesions per patient will be selected for radiomics and biopsy. Both lesions will be assessed for [18F]F AraG uptake before and after CkIT. Only one lesion will be biopsied twice (once before and once after CkIT treatment close to the time of imaging), and the other lesion will not be manipulated and used as a control.

There will be a pre therapy scan [18F]F AraG which will be administered anytime within a 14 day period prior to the initial Day 1 CkIT administration. There will also be a post therapy scan which will be performed within 3 to 6 weeks after the initial CkIT dose. The timing of the second [18F]F AraG scans may be altered based on preliminary results from the initial patient scan results, and could be obtained during the first 2 weeks after initiation of therapy.

The investigators will compare the [18F]F AraG activity (based on development of tumoral volumes of interest (VOIs) pre and post CkIT in both lesions.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor with planned CkIT
* Must be >18 years old
* Signed Informed Consent Form
* Patient must have two qualifying lesions

Exclusion Criteria:

* Patient is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Correlate change in [18F]F AraG signal following CkIT therapy with change in level of T cell infiltration in tumor biopsies | 24 Months
  Pre and post CkIT biopsies of the same tumor lesion will be performed an analyze T-cell tumor infiltration, this will be correlated to [18F]F-AraG PET signal.

SECONDARY OUTCOMES:
1. Correlate change in [18F]F AraG uptake signal in tumor lesions with clinical benefit rate (defined as Complete Response (CR) + Partial Response (PR) + stable disease (SD) > 4 months) using iRECIST criteria | 24 Months
2. Correlate change in [18F]F AraG signal in lung and GI tract with the occurrence of Grade 3 or 4 immune related adverse events. | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Carina Mari Aparici, M.D., Principal Investigator — Stanford University; Erik Mittra, M.D., Principal Investigator — Oregon Health and Science University; Shivaani Kummar, M.D., Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No